CLINICAL TRIAL: NCT02750982
Title: A Single-Arm Prospective Investigation of the Effects of Laughter Therapy on Mood, Stress, and Self-Efficacy in People With Central Nervous System Disorders.
Brief Title: Laughter Therapy Effects on Mood, Stress and Self-efficacy in People With Neurological Diseases.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown, Theodore R., M.D., MPH (Individual)
Responsible Party: Principal Investigator, Theodore R Brown, M.D., MPH, Brown, Theodore R., M.D., MPH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TRBROWN201601
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Alzheimer's Disease; Amyotrophic Lateral Sclerosis; Brain Injury; Huntington's Disease; Multiple Sclerosis; Parkinson's Disease; Stroke; Spinal Cord Injury
MeSH Terms: conditions — Alzheimer Disease; Amyotrophic Lateral Sclerosis; Brain Injuries; Huntington Disease; Multiple Sclerosis; Parkinson Disease; Stroke; Spinal Cord Injuries | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laughter therapy (Experimental): effects of Laughter therapy (LT) on mood, self-efficacy and other wellness measures in people with neurological conditions.
  Interventions: Other: Laughter Therapy

INTERVENTIONS:
Other: Laughter Therapy — Laughter Therapy (LT) involves simple exercises using playfulness, eye contact and chanting in forms of laughter. LT will be taught by a certified LT instructor in a group session. There will be 8 sessions per group with each session attended by 8-12 participants and lasting 60 minutes

SUMMARY:
This is a prospective investigation of the effects of Laughter therapy (LT) on perceived stress, self-efficacy, mood and other wellness measures in people with the following neurological conditions: Alzheimer's disease, amyotrophic lateral sclerosis, brain injury, Huntington's Disease, multiple sclerosis, Parkinson's Disease, post-stroke, spinal cord injury.

DETAILED DESCRIPTION:
Laughter therapy (LT) has potential benefits in treating illness. It combines laughter with breathing and body exercises to stimulate laughter, both real and artificial, in a group setting. Laughter therapy may help treating illness by strengthening breathing muscles, improving mood, and providing pain and stress relief. EvergreenHealth has presented laughter therapy classes to patients with Parkinson's disease and Multiple sclerosis and other neurological conditions. The therapy will be led by a certified laughter therapist and mental health professional.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis based on medical record review of one of the following neurological diseases: Alzheimer's disease, amyotrophic lateral sclerosis, brain injury, Huntington's Disease, Multiple Sclerosis, Parkinson's Disease, Post-Stroke, Spinal Cord Injury.
* Medically stable for at least 2 months.
* Not participating in Laughter therapy for 30 days prior to screening.

Exclusion Criteria:

* Females who are pregnant
* Any unstable medical condition
* Severe cognitive deficits that would interfere with participation (e.g. unable to follow commands).
* Severe abdominal pain, chest pain or back pain.
* Abdominal, chest or back surgery within 90 days.
* Psychosis or severe mental illness.
* Untreated hernia.
* Persistent cough.
* Advanced hemorrhoids.
* Epilepsy.
* Uncontrolled Hypertension - SBP >170 or DBP >105.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9, for depression) | Change from Baseline to 8 weeks
  Outcome measures will be completed at baseline, active-phase completion at week 8 and post-active phase week 8 (16 weeks post-start of active phase).
Generalized Anxiety Disorder 7-item scale (GAD-7, for anxiety) | Change from Baseline to 8 weeks
  Outcome measures will be completed at baseline, active-phase completion at week 8 and post-active phase week 8 (16 weeks post-start of active phase).

SECONDARY OUTCOMES:
The General Self-Efficacy Scale (GSE) | Change from Baseline to 8 weeks
  Outcome measures will be completed at baseline, active-phase completion at week 8 and post-active phase week 8 (16 weeks post-start of active phase).

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Brown, MD, MPH, Principal Investigator — Evergreen Healthcare
Locations (1):
- Evergreen Healthcare, Kirkland, Washington, United States

IPD SHARING:
Plan to Share IPD: No